CLINICAL TRIAL: NCT00733161
Title: Effect of Passive Exercise on Systemic Endothelial Function in Elderly Patients With Chronic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University (Other)
Responsible Party: Principal Investigator, Takeshi Morimoto, Investigator, Kyoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20795203
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Congestive Heart Failure; Endothelium-derived Factors; Elderly
Keywords: passive leg exercise; congestive heart failure; endothelium-derived factors; elderly
MeSH Terms: conditions — Heart Failure | interventions — Resistance Training

ARMS (2):
- 1 (Active Comparator): Passive leg cycle exercise with stretching and resistance training
  Interventions: Other: Passive leg cycle exercise with stretching and resistance training
- 2 (Active Comparator): Stretching and resistance training
  Interventions: Other: Stretching and resistance training

INTERVENTIONS:
Other: Passive leg cycle exercise with stretching and resistance training — Passive leg cycle exercise for 15 minutes everyday as well as stretching and resistance training
  Arms: 1
Other: Stretching and resistance training — Stretching and resistance training everyday but no Passive leg cycle exercise
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of passive exercise on systemic endothelial function in elderly patients with chronic heart failure.

DETAILED DESCRIPTION:
Endothelial function is known to be impaired in patients with chronic heart failure (CHF) and impaired endothelial function has been reported to be associated with an increased mortality risk in those subjects. Although systemic exercise training has been demonstrated to improve endothelial dysfunction in patients with CHF, elderly patients with severely impaired exercise capacity could not engaged in usual exercise training using ordinal ergometer. Those patients are able to join stretching or very light resistance training. On the other hand, passive pedaling using strength ergometer has been reported to be useful in patients with severely impaired exercise capacity, but the safety and the efficacy of passive pedaling on endothelial function in old patients with CHF has not been previously reported.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic heart failure
* Elderly patients aged ≧65 years
* Patients with severely reduced exercise capacity and cannot continue exercise with usual cycling ergometer for 5 minutes

Exclusion Criteria:

* Unstable hemodynamic status (uncontrolled arrhythmia, uncontrolled congestion, uncontrolled hypertension)
* Active infectious disease
* Malignancy
* Chronic obstructive pulmonary disease
* Dialysis
* Severe aortic valve disease
* With any hip, knee, ankle joint pain
* Hemiplegia
* Current smoker

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 2 weeks

SECONDARY OUTCOMES:
Left ventricular systolic and diastolic function | 2 weeks
Six-minute walk distance | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Principal Investigator — Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine, Kyoto, Japan

REFERENCES:
- [Derived] Ozasa N, Morimoto T, Bao B, Shioi T, Kimura T. Effects of machine-assisted cycling on exercise capacity and endothelial function in elderly patients with heart failure. Circ J. 2012;76(8):1889-94. doi: 10.1253/circj.cj-11-1113. Epub 2012 May 16. PMID 22664754